CLINICAL TRIAL: NCT04207853
Title: Immediate Effect of Whole Body Vibration on Skin Temperature, Circulation, Peripheral Sensitivity and Plantar Pressure in Adults and Elderly With and Without Type 2 Diabetes: Controlled Clinical Trial
Brief Title: Immediate Effect of Whole Body Vibration on Diabetics and Non-diabetics
Acronym: DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, Doutor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Immediate, Vibration and DM
Record Dates: First submitted 2019-10-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Skin Temperature; Circulation; Peripheral Sensitivity; Plantar Pressure; Vibration
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 6 groups: whole body vibration in diabetics (G1), the sham vibration group in diabetics (G2) and diabetic control group (G3), the whole body vibration group in non-diabetics (G4), the vibration group " sham "in non-diabetics (G5) and non-diabetic control group (G6), establishing a single treatment session for G1, G2, G4 and G5.
Who Masked: Participant, Care Provider, Investigator
Masking Description: group the patient will enter. The patient will be allocated among three groups. After the final evaluations, all data will be analyzed by another researcher directed solely to that purpose. Therefore, there will be a triple blinding (researcher, patient and statistician).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- whole body vibration in diabetics (G1) (Experimental): One 24Hz session, 4mm amplitude, 8 rep series, 45s intervention time, 30s recovery
  Interventions: Other: whole body vibration em DM
- the sham vibration group in diabetics (G2) (Sham Comparator): dummy vibration (sound stimulus), 8-rep series, 45s intervention time, 30s recovery
  Interventions: Other: Vibration "sham" em DM
- diabetic control group (G3) (No Intervention): no treatment
- whole body vibration group in non-diabetics (G4) (Active Comparator): One 24Hz session, 4mm amplitude, 8 rep series, 45s intervention time, 30s recovery
  Interventions: Other: whole body vibration em NDM
- the vibration group " sham "in non-diabetics (G5) (Sham Comparator): dummy vibration (sound stimulus), 8-rep series, 45s intervention time, 30s recovery
  Interventions: Other: Vibration "sham" em NDM
- non-diabetic control group (G6) (No Intervention): no treatment

INTERVENTIONS:
Other: whole body vibration em DM — The vibrating platform is a new biophysical modality of exercise. The individual exercises on a plate that oscillates up and down movements at a specific frequency and amplitude, and the exercises are performed static and / or dynamic. Vibration is supposed to activate muscle spindles and evoke contractions, which are induced by the complex spinal and supraspinal neurophysiological mechanism known as the tonic vibration reflex.
  Arms: whole body vibration in diabetics (G1)
Other: Vibration "sham" em DM — Sham vibration will be performed with the platform disconnected. A sound device will be connected producing a noise similar to the connected platform for a time equivalent to the treatment protocol, as it will not be possible to visibly distinguish the vibratory stimulus. Participants who will undergo false vibration will not have contact with those who will perform the protocol effectively.
  Arms: the sham vibration group in diabetics (G2)
Other: whole body vibration em NDM — The vibrating platform is a new biophysical modality of exercise. The individual exercises on a plate that oscillates up and down movements at a specific frequency and amplitude, and the exercises are performed static and / or dynamic. Vibration is supposed to activate muscle spindles and evoke contractions, which are induced by the complex spinal and supraspinal neurophysiological mechanism known as the tonic vibration reflex.
  Arms: whole body vibration group in non-diabetics (G4)
Other: Vibration "sham" em NDM — Sham vibration will be performed with the platform disconnected. A sound device will be connected producing a noise similar to the connected platform for a time equivalent to the treatment protocol, as it will not be possible to visibly distinguish the vibratory stimulus. Participants who will undergo false vibration will not have contact with those who will perform the protocol effectively.
  Arms: the vibration group " sham "in non-diabetics (G5)

SUMMARY:
Introduction: Diabetes Mellitus (DM) is an important health condition of the population and its prevalence continues to grow due to population aging, economic development and urbanization. The exercise is an important factor of prevention and control, thereby decreasing the risk of metabolic diseases, cardiovascular diseases and improving the functionality of the patient with diabetes.

Objective: Evaluate the response of resistance training associated with wholebody vibration on peripheral circulation and functional performance of elderly with type 2 diabetes. Methods: This is a clinical trial study, controlled, randomized and blinded, which will follow the guidelines established by the Consolidated Standards of Reporting Trials (CONSORT). Patients will be recruited in the light of the eligibility criteria and randomly divided into 3 groups: resistance training associated with whole body vibration (G1), resistance training associated with vibration sham (G2) and control group-guidelines about foot care (GC), establishing 36 treatment sessions, three times a week for the G1 and G2.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is an important health condition of the population and its prevalence continues to grow due to population aging, economic development and urbanization. Exercise is an important factor of prevention and metabolic control, thus reducing the risk of cardiovascular disease and improving the functionality of the patient with diabetes. The vibrating platform is a new biophysical modality of exercise. The individual exercises on a plate that oscillates up and down movements at a specific frequency and amplitude, and the exercises are performed static and / or dynamic. The present study aims to evaluate the immediate effect of whole body vibration on skin temperature, circulation, peripheral sensitivity and plantar pressure in adults and older adults with and without type 2 diabetes. controlled, randomized and blind, which will follow the guidelines set forth in the Consolidated Standards of Reporting Trials (CONSORT). It will be held at the Laboratory of Kinesiotherapy and Manual Therapeutic Resources (LACIRTEM) of the Department of Physical Therapy of the Federal University of Pernambuco (UFPE), in 2019. Patients will be recruited meeting the eligibility criteria and randomly assigned to 6 groups: whole body vibration in diabetics (G1), the sham vibration group in diabetics (G2) and diabetic control group (G3), the whole body vibration group in non-diabetics (G4), the vibration group " sham "in non-diabetics (G5) and non-diabetic control group (G6), establishing a single treatment session for G1, G2, G4 and G5. The control group of diabetics and non-diabetics will be evaluated, will receive pamphlets and guidelines on diabetes, will answer the research questionnaires and will be reassessed. This study will be submitted to the UFPE Human Research Ethics Committee and collection will only begin after its approval. All individuals must have read and signed the Informed Consent Form, authorizing their participation. The study is in line with National Health Council Resolution 466/12 and the Declaration of Helsinki. For statistical analysis of the results will be assigned a significance level of 95%, performed using the statistical software SPSS version 23.0. Whole body vibration is expected to show more significant improvements than sham and control groups in the outcomes studied.

ELIGIBILITY:
Inclusion Criteria:

(I) Diabetics classified clinically as type 2 diagnosed more than 2 years and less than 20 years of diagnosis; (II) Patients of both sexes aged between 45 and 80 years; (III) Be functionally independent; (IV) Possess cognitive ability to answer and perform the exercises evaluated by the Mini-Mental State Examination (MMSE); (V) Patients without severe foot deformities requiring therapeutic footwear; (VI) Not having orthopedic disabilities; (VII) No indications of deep vein thrombosis; (VIII) Not making use of mobility aids (IX) Presenting BMI between 18.50 and 34.99kg / m2; (X) For the control group participants must fulfill all of the above requirements except item I.

Exclusion Criteria:

(I) Type I diabetics; (II) Diabetics and non-diabetics who are performing physical activity or who have performed any type of physical activity less than 2 months; (III) Have lower limb amputation; (IV) Patients with vertigo or labyrinthitis; (V) Have blood pressure greater than or equal to 150/100 mmHg or less than or equal to 60/40 mmHg.

(VI) Presence of rheumatic diseases; (VII) Chemical dependents; (VIII) Blood glucose greater than 300mg/dL.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
skin temperature | " until study completion, an average of 2 months".
  Infrared Thermography (TI)
circulation | " until study completion, an average of 2 months".
  Vascular Doppler ultrasound (UVD)
peripheral sensitivity | " until study completion, an average of 2 months".
  Esthesiometer
plantar pressure | " until study completion, an average of 2 months".
  Baropodometry

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No